CLINICAL TRIAL: NCT02799316
Title: Is Hepatitis B Surface Antigen (HB s Ag) Enough Alone as a Screening Test for Hepatitis B Virus Infection in Rheumatic Disease Patients Before Starting Immunosuppressive Therapies??
Brief Title: Is Hepatitis B Surface Antigen (HB s Ag) Enough Alone as a Screening Test Before Immunosuppressive Therapies?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Consultant liver and GIT diseases- Tanta university hospital, Tanta University
Organization: Tanta University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Rasha Abdelno
Record Dates: First submitted 2016-06-10; First posted 2016-06-14 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rheumatic disease with HBs-ag positive (Other): • HBV core antibodies testing. • Real time PCR testing.
  Interventions: Other: HBV core antibodies testing. • Real time PCR testing.

INTERVENTIONS:
Other: HBV core antibodies testing. • Real time PCR testing. — * HBV core antibodies testing in HBV surface antigen negative patients.
  * Real time PCR testing for those having positive HBc antibodies.

SUMMARY:
Hepatitis B virus (HBV) infection is a challenging health problem. According to the World Health Organization, an estimated 240 million individuals (3.7%) suffered from chronic HBV infection worldwide.

After acute hepatitis B virus (HBV) infection, the disappearance of hepatitis B surface antigen (HBsAg) had generally been believed to signify viral elimination. However, it now becomes clear that those subjects may have occult HBV infection which is defined as the presence of HBV DNA in the liver in the absence of HBsAg in the serum. Occult HBV infection usually accompanies antibody against hepatitis B core antigen (anti-HBc) and/or antibody against HBsAg (anti-HBs), but some cases might not have these serological markers (seronegative occult HBV infection) .

DETAILED DESCRIPTION:
In a recent systematic review, nearly 40% of HBsAg carriers and 5% of antiHBc-positive but HBsAg-negative patients developed HBVr during TNF inhibitor therapy.

Considering the lifelong use of multiple antirheumatic drugs, we need more specific guidelines for the management of rheumatic disease patients who are scheduled to receive biological and/or non-biological DMARDs.

ELIGIBILITY:
Inclusion Criteria:

* • Any patients with rheumatic disease with hepatitis B surface antigen negative.

Exclusion Criteria:

* • Overt co-morbid condition.

  * Any malignancy e.g. HCC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with occult HBV. | 1 year
  Number of patients having occult HBV.

CONTACTS AND LOCATIONS:
Overall Officials: Rasha A Abdel Noor, Consultant, Principal Investigator — Internal medicine department - Tanta university; Sherief Abd-Elsalam, Consultant, Study Chair — Division of Gastroenterology and Hepatology- Tanta; Walaa Elkhalawany, Consultant, Study Chair — liver diseases dept.-Tanta university hospital; Mona Watani, Consultant, Study Chair — liver diseases dept.-Tanta university hospital; Rehab Badawi, Consultant, Study Chair — liver diseases dept.-Tanta university hospital
Locations (1):
- Sherief Abd-Elsalam, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided